CLINICAL TRIAL: NCT00770991
Title: A Pilot Study To Investigate the Biological Modulation of Familial Adenomatous Polyposis (FAP) by Lyophilized Black Raspberries
Brief Title: Lyophilized Black Raspberries in Adults With Familial Adenomatous Polyposis (FAP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Carol Burke, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003-34501-13965
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Polyp, Familial Adenomatous Polyposis, Prevention
MeSH Terms: conditions — Adenomatous Polyposis Coli; Polyps | interventions — Suppositories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black Raspberry (BRB) Slurry plus BRB suppositories (Experimental): 20 grams BRB Slurry BID plus two, 730 mg BRB suppositories HS
  Interventions: Drug: Black raspberry (BRB) Slurry; Drug: Black Raspberry (BRB) Suppositories
- Black Raspberry (BRB) Placebo Slurry plus BRB suppositories (Experimental): 20 grams BRB Placebo Slurry BID plus two, 730 mg BRB suppositories HS
  Interventions: Drug: Black Raspberry (BRB) Suppositories; Drug: Black Raspberry (BRB) Placebo Slurry

INTERVENTIONS:
Drug: Black raspberry (BRB) Slurry — 20 grams BRB Slurry
  Arms: Black Raspberry (BRB) Slurry plus BRB suppositories
Drug: Black Raspberry (BRB) Suppositories — Two, 730 mg BRB suppositories QHS
Drug: Black Raspberry (BRB) Placebo Slurry — 20 grams BRB placebo slurry
  Arms: Black Raspberry (BRB) Placebo Slurry plus BRB suppositories

SUMMARY:
This is a 36 week dietary intervention pilot study to evaluate the effects of lyophilized black raspberries on rectal polyp burden and biomarkers in subjects with FAP. Subjects will undergo a colonoscopy or sigmoidoscopy before study treatment to determine eligibility for the study. Eligible participants will undergo a sigmoidoscopy at 36 weeks after the initiation of study treatment. The size and number of rectal polyps will be documented on a code sheet and by photograph. The efficacy outcome will include the percentage reduction in the number of rectal polyps between baseline and 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial adenomatous polyposis with at least 5 rectal polyps which are greater than or equal to 2 mm on baseline colonoscopy
* Have an endoscopically assessable rectal segment
* Have not taken NSAIDs or selective COX-2 inhibitors for two months prior to the study and willing to remain off NSAIDs for the study duration.

Exclusion Criteria:

* Known allergies or hypersensitivity to berries
* Diabetes mellitus
* Subjects taking NSAIDs or COX-2 inhibitors who cannot be taken off the medication due to their clinical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Burke, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open for enrollment at Cleveland Clinic from December 9, 2005 to March 26, 2008. Subjects with FAP who had an assessable rectal segment were screened for potential eligibility. Once it was determined the subjects were potentially eligible they were contacted by phone or letter.
Pre-assignment Details: After potentially eligible subjects signed the informed consent, a physical examination with medical history and colonoscopy or sigmoidoscopy was performed as indicated. Blood and urine samples were collected. Subjects with adequate rectal polyp burden and laboratory results within study guidelines were eligible to be randomized.
Groups:
- Placebo Powder Plus 2 Berry Suppositories: 20 gram placebo powder administered as an oral slurry three times a day, plus 2 730 mg berry suppositories administered at bedtime. Each berry suppository contained 730 mg black raspberries.
- Black Raspberry Slurry Plus 2 Berry Suppositories: 20 grams of lyophilized berry powder administered as an oral slurry three times a day, plus 2 730 mg berry suppositories administered at bedtime. Each suppository contained 730 mg black raspberries.
Period: Overall Study
Arm/Group | Placebo Powder Plus 2 Berry Suppositories | Black Raspberry Slurry Plus 2 Berry Suppositories
Started | 12 (34 participants enrolled (signed informed consent). 24 subjects were eligible to be randomized.) | 12 (We anticipated 26-30 subjects with FAP 18 year or olders would need to be enrolled to randomize 18)
Completed | 7 (7 subjects completed 36 weeks (+/- 10 days)of treatment) | 7 (7 subjects completed 36 weeks (+/- 10 days)of treatment)
Not Completed | 5 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 5
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Two Berry Suppositories Bedtime Plus Oral Berry Powder: 20 g of lyophilized berry powder administered orally 3 times per day, plus 2 berry suppositories administered at bedtime. Each suppository contains 730 mg Black Raspberries
- Two Berry Suppositories Bedtime Plus Placebo Powder: 20 g of placebo powder administered as an oral slurry 3 times per day, plus 2 berry suppositories administered at bedtime. Each suppository contains 730 mg Black Raspberries
- Total: Total of all reporting groups
Arm/Group | Two Berry Suppositories Bedtime Plus Oral Berry Powder | Two Berry Suppositories Bedtime Plus Placebo Powder | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study in Number of Rectal Polyps
Time Frame: Baseline and 36 weeks
Measure: Mean (Standard Deviation); unit: polyps
Groups:
- Lyophilized Black Raspberry (BRB) Suppositories Plus Placebo: Two, 730 mg BRB suppositories administered at bedtime plus 20 grams placebo slurry .
- Lypholized BRB Suppositiry Plus BRB Slurry: 2 lyphilized black raspberry suppositories plus black raspberry slurry.
Arm/Group | Lyophilized Black Raspberry (BRB) Suppositories Plus Placebo | Lypholized BRB Suppositiry Plus BRB Slurry | All Participants
Number analyzed (Participants) | 7 | 7 | 14
polyps | -5.4 (5.3) | -1.6 (9.2) | -3.5 (7.5)
Statistical Analysis 1: Comparison: All Participants; All patients received BRB suppositories and were pooled for the analysis comparing baseline and end of study polyp counts; Test type: Superiority or Other; p = 0.065, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Apoptosis and Cell Proliferation Measured by Percent Difference in Staining.
Description: A pooled analysis of all participants was used for biomarker results. Tissue from normal mucosa and rectal polyps were obtained to assay KI 67 (proliferation) and TUNEL at baseline and end of treatment. A decrease in the value of KI 67 implies lower proliferation while an increase in TUNEL is suggestive of an increase in apoptosis.
Time Frame: baseline and 36 weeks
Measure: Mean (Standard Deviation); unit: percentage of brown staining of cells
Groups:
- Normal Mucosa: all participants combined for this analysis. Sample of normal mucosa
- Polyp: all participants used for this analysis
Arm/Group | Normal Mucosa | Polyp
Number analyzed (Participants) | 14 | 14
percentage of brown staining of cells
  KI 67 assay at baseline | 11.3 (1.14) | 55.2 (2.81)
  KI 67 at 36 weeks | 8.00 (1.07) | 49.12 (2.28)
  Difference in means of KI 67 | -3.30 (1.23) | -6.08 (1.83)
  Tunel assay at baseline | 0.58 (0.10) | 4.49 (0.95)
  Tunel assay at 36 weeks | 1.08 (0.33) | 7.64 (1.17)
  Difference in mean of Tunel | 0.50 (0.33) | 3.15 (1.20)
Statistical Analysis 1: Comparison: Normal Mucosa; Test type: Superiority or Other; p = 0.016, Chi-squared

3. Primary Outcome: Change in Burden of Rectal Polyps
Description: The burden was measured as the sum of the number of polyps x size of polyps in mm. The change in burden was determined between baseline and 36 weeks.
Time Frame: Baseline and 36 weeks
Measure: Mean (Standard Deviation); unit: polyp number x mm
Groups:
- Lyophilized Black Raspberry (BRB) Suppositories + Placebo: Two, 730 mg BRB suppositories administered at bedtime.
Arm/Group | Lyophilized Black Raspberry (BRB) Suppositories + Placebo | Lyophilized BRB Suppositories + BRB Slurry | All Participants
Number analyzed (Participants) | 7 | 7 | 14
polyp number x mm | -13 (11.7) | -5.7 (26.6) | -9.4 (20.1)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.043, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting day first dose study agent taken to end of study visit at 36 weeks. Subjects contacted at monthly intervals for AE evaluation.
Description: Subjects asked to complete diary to record date and time study agent consumed, time suppository inserted, changes in their health, visits to any physician, changes in medications and overnight hospitalizations. If a subject experienced more than 1 of a given AE, subject is counted only once for that AE.
Groups:
- Black Raspberry Placebo Slurry Plus 2 Berry Suppositories: 20 gram placebo powder administered as an oral slurry three times a day, plus 2 730 mg berry suppositories administered at bedtime. Each berry suppository contained 730 mg black raspberries.
Arm/Group | Black Raspberry Placebo Slurry Plus 2 Berry Suppositories | Black Raspberry Slurry Plus 2 Berry Suppositories
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 7/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Black Raspberry Placebo Slurry Plus 2 Berry Suppositories (N=12) | Black Raspberry Slurry Plus 2 Berry Suppositories (N=12)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Black Raspberry Placebo Slurry Plus 2 Berry Suppositories (N=12) | Black Raspberry Slurry Plus 2 Berry Suppositories (N=12)
Abdominal bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Increased appetite (General disorders) | 0 (0) | 1 (1)
Flatulance (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Elevated ALT and AST (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 4 (4) | 5 (5)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cramping in extremities (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No